CLINICAL TRIAL: NCT02177344
Title: A Six Month, Randomized, Double-blind (Within Formulation), Multiple Dose Trial to Compare the Safety and Efficacy of 20 mcg and 40 mcg of Ipratropium Bromide, as Delivered by the RESPIMAT Device, to 18 mcg ATROVENT® Inhalation Aerosol (x 2 Puffs) and Respective Placebos in Adults, With Chronic Obstructive Pulmonary Disease
Brief Title: Safety and Efficacy of Two Different Doses of Ipratropium Bromide Versus ATROVENT® Inhalation Aerosol in Adults With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 244.2484
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium

ARMS (4):
- Low dose of ipratropium bromide (Experimental)
  Interventions: Drug: Low dose of Ipratropium bromide
- High dose of Ipratopium bromide (Experimental)
  Interventions: Drug: High dose of Ipratropium bromide
- Atrovent (Active Comparator)
  Interventions: Drug: Atrovent
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose of Ipratropium bromide — One puff, 4 times daily by oral inhalation
  Arms: Low dose of ipratropium bromide
Drug: High dose of Ipratropium bromide — One puff, 4 times daily by oral inhalation
  Arms: High dose of Ipratopium bromide
Drug: Atrovent — Two puffs, 4 times daily by oral inhalation
  Arms: Atrovent
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to confirm that chronic dosing of 20 mcg and 40 mcg of ipratropium bromide, administered via the RESPIMAT device, demonstrates clinical comparability and similar safety profiles to the 36 mcg dose of ATROVENT® Inhalation Aerosol (containing chlorinated fluorocarbons (CFC)) in patients with chronic obstructive pulmonary disease (COPD). The efficacy and safety profiles of the two doses administered via the RESPIMAT device will also be compared to their respective placebo groups

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have a diagnosis of COPD and must meet the following spirometric criteria:

   * Patients must have relatively stable, moderate to severe airway obstruction with a FEV1 =< 65% of predicted normal and FEV1 =< 70% of FVC
2. Male or female patients 40 years of age or older
3. Patients must have a smoking history of more than ten packs-years. A pack-year is defined as the equivalent of smoking one pack of 20 cigarettes per day for a year
4. Patients must be able to perform pulmonary function tests and maintain records during the study period, as required in the protocol
5. Patients must be able to be trained in the proper use of an inhalation aerosol and the Respimat device
6. All patients must sign an Informed Consent Form prior to participation in the trial i.e., at least 24 hours prior to screening (Visit 1)

Exclusion Criteria:

1. Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease, which in the opinion of the investigator, may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
2. Patients with clinically relevant abnormal baseline haematology, blood chemistry or urinalysis. If the abnormality defines a disease listed as an exclusion criterion, the patient is excluded
3. All patients with a serum glutamate oxaloacetate transaminase > 80 U/L, serum glutamate pyruvate transaminase > 80 U/L, bilirubin > 34.2 µmol/L or creatinine > 176.8 µmol/L will be excluded regardless of the clinical condition. Repeat laboratory evaluation will not be conducted in these subjects
4. Patients who have a blood eosinophil count >= 0.6 GI/L. A repeat eosinophil count will not be conducted in these patients
5. Patients with a recent history (i.e., one year or less) of myocardial infarction
6. Patients with a recent history (i.e., three years or less) of heart failure or patients with any cardiac arrhythmia requiring drug therapy
7. Patients with a history of cancer, other than treated basal cell carcinoma, within the last five years
8. Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis
9. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of a thoracotomy for other reasons should be evaluated as per exclusion criterion #1
10. Patients with a history of asthma, allergic rhinitis or atopy
11. Patients with a history of and/or active alcohol or drug abuse
12. Patients with known active tuberculosis
13. Patients with an upper respiratory tract infection or COPD exacerbation in the past six weeks prior to the Screening Visit (Visit 1) or during the baseline period
14. Patients with known symptomatic prostatic hypertrophy, bladder neck obstruction, or urinary retention
15. Patients with known narrow-angle glaucoma, or raised intra-ocular pressure
16. Patients with current significant psychiatric disorders
17. Patients with regular use of daytime oxygen therapy
18. Patients who are being treated with cromolyn sodium or nedocromil sodium
19. Patients who are being treated with antihistamines
20. Patients using oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at a dose in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day
21. Patients who are being treated with beta-blocker medication
22. Patients who have had changes in their therapeutic plan within the last six weeks prior to the Screening Visit (Visit 1)
23. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e., oral contraceptives, intrauterine devices or diaphragm with spermicide, or Norplant®)
24. Patients with known hypersensitivity to anticholinergic drugs or any other components of the ATROVENT® Solution including Benzalkonium chloride and Edetic acid
25. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening Visit (Visit 1)
26. Previous participation in this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 1998-08; Primary Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
Area under the curve from 0 to 6 hours (AUC0-6) for average of forced expiratory volume in 1 second (FEV1) | up to day 169

SECONDARY OUTCOMES:
Peak FEV1 post treatment | up to day 169
Onset of therapeutic FEV1 response | up to day 169
Duration of therapeutic FEV1 response | up to day 169
Time to peak FEV1 response | up to day 169
Total area under the curve from 0 to 6 hours (TAUC0-6) for average FEV1 response | up to day 169
Average change in forced vital capacity (FVC) from zero to six hours | up to day 169
Peak FVC post treatment | up to day 169
Peak expiratory flow rate (PEFR) measured by the patient at home two times daily | up to day 169
Amount of inhaled rescue medication used during the treatment period | up to day 169
Concomitant medication usage during the treatment period including steroids | up to day 169
Change in patient daily symptom assessments | Baseline, up to day 169
Number of patients with adverse events | Up to day 169
Changes in vital signs (pulse rate, blood pressure) | Baseline, up to day 169
Changes in laboratory tests | Baseline, day 169
Number of patients with significant changes in ECG (electrocardiogram) | Baseline, day 169
Changes in physical examination | Baseline, day 169